CLINICAL TRIAL: NCT00575042
Title: Pilot Study of Fenofibrate for Primary Biliary Cirrhosis
Brief Title: Use of Fenofibrate for Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The PBCers Organization (Other); Shionogi Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 405-2006
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2012-01-09 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Primary Biliary Cirrhosis
Keywords: PBC; Primary Biliary Cirrhosis; Fenofibrate; Triglide
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients treated with Fenofibrate (Experimental): Fenofibrate IDD-P (Insoluble Drug Delivery-Micro Particle) 160 mg table per day for 1 year
  Interventions: Drug: Fenofibrate IDD-P (Insoluble Drug Delivery-Micro Particle)

INTERVENTIONS:
Drug: Fenofibrate IDD-P (Insoluble Drug Delivery-Micro Particle) — 160 mg per day for 1 year
  Other Names: Triglide-Insoluble Drug Delivery-Micro Particle Fenofibrate (IDD-P)

SUMMARY:
This is a pilot study to evaluate the safety and efficacy of fenofibrate on patients with primary biliary cirrhosis who have an incomplete response to ursodeoxycholic acid.

DETAILED DESCRIPTION:
This is a multicenter open label pilot study to evaluate the efficacy of fenofibrate in 20 patients with PBC treated for 1 year. A randomized design would not be feasible at this stage of the research. Two sites are enrolling patients: University of Florida, Gainesville, and Mayo Clinic Rochester, with the first as the coordinating site. The total number of patients to start treatment will not exceed 20. Our endpoints are 1) surrogate markers of disease activity -serum alkaline phosphatase and immunoglobulin M; 2) a well validated prognostic index -Mayo risk score and 3) the NIDDK quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of PBC by serological (positive antimitochondrial antibodies) and/or histological evidence (diagnostic liver biopsy)
* Previous treatment with UDCA 13-15 mg/kg/day for at least 1 year
* Persistent elevation of serum alkaline phosphatase ≥ 2 times the upper limit of normal on two separate measurements
* Female patients of childbearing age should have a pregnancy test done within -days of the beginning of this trial, and should agree to be on adequate contraception throughout the study period
* Signed informed consent after careful review of the information and study details by one of the investigators

Exclusion Criteria

* Hypersensitivity to fenofibrate
* Prisoners and institutionalized subjects
* Pregnant or nursing women
* Anticipated need for liver transplantation in one year (estimated one year survival < 80%) as determined by the Mayo risk score. The Mayo risk score takes into account the patient's age, serum bilirubin, albumin and prothrombin time, as well as presence or absence of peripheral edema.
* Recipients of liver transplantation
* Recurrent variceal hemorrhage, uncontrolled encephalopathy or refractory ascites
* Co-existing liver diseases, such as primary sclerosing cholangitis, acute or chronic hepatitis, alcoholic liver disease, choledocholithiasis, autoimmune hepatitis, cholangiocarcinoma
* Acute or chronic renal failure
* Known history of cholecystitis with intact gallbladder
* Current use of statins, as the concomitant use of fibrates and statins would increase the risk of toxicity

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Levy, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Background] Levy C, Peter J, Keach J, Petz J, Lindor KD, Cabrera R, et al. Fenofibrate improves liver biochemistries in primary biliary cirrhosis. Hepatology. 2009;50(4 (suppl)):995A.
- [Result] Levy C, Peter JA, Nelson DR, Keach J, Petz J, Cabrera R, Clark V, Firpi RJ, Morelli G, Soldevila-Pico C, Lindor K. Pilot study: fenofibrate for patients with primary biliary cirrhosis and an incomplete response to ursodeoxycholic acid. Aliment Pharmacol Ther. 2011 Jan;33(2):235-42. doi: 10.1111/j.1365-2036.2010.04512.x. Epub 2010 Nov 17. PMID 21083674

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the liver clinics at University of Florida and Mayo Clinic Rochester.
Groups:
- Fenofibrate 160 mg Per Day: Fenofibrate (Insoluble Drug Deliver-Micro Particle Fenofibrate (IDD-P)) 160 mg per day
Period: Overall Study
Arm/Group | Fenofibrate 160 mg Per Day
Started | 20
Completed | 17 (2 with side effects and 1 lost to follow-up)
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Patients Treated With Fenofibrate: Fenofibrate IDD-P (Insoluble Drug Delivery-Micro Particle) 160 mg per day
Arm/Group | Patients Treated With Fenofibrate
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Serum Level of Alkaline Phosphatase
Description: We analyzed whether there was a difference in median ALP at 1 year compared to baseline values.
Time Frame: 1 year
Measure: Median (Full Range); unit: U/L
Groups:
- Patients Before Treatment With Fenofibrate: Patients with previous incomplete response to UDCA
- Patients Treated With Fenofibrate: Fenofibrate IDD-P (Insoluble Drug Delivery-Micro Particle)
Arm/Group | Patients Before Treatment With Fenofibrate | Patients Treated With Fenofibrate
Number analyzed (Participants) | 20 | 17
U/L | 351 [214 to 779] | 175 [60 to 384]
Statistical Analysis 1: Comparison: Patients Before Treatment With Fenofibrate vs Patients Treated With Fenofibrate; Sample size calculation estimated that with 20 patients, and assuming a 10% drop-out rate, the study would have 80% power to detect a response rate in 35% or more of the study patients. A two-sided p value<0.05 was considered statistically significant; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 15 months
Arm/Group | Patients Treated With Fenofibrate
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With Fenofibrate (N=20)
heartburn (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With Fenofibrate (N=20)
heartburn (Gastrointestinal disorders) | 4 (4)
nausea (Gastrointestinal disorders) | 2 (2)
transient elevation of transaminases (Hepatobiliary disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
A major limitation is the uncontrolled nature of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No